**Emory University IRB** IRB use only

Study No.: IRB00081580 Document Approved On: 9/27/2016

> Title: Allocation System Changes for Equity in kidNey Transplantation (ASCENT) Study NCT # NCT02879812 Date: 9/27/2016

### Study No.: IRB00081580

Document Approved On: 9/27/2016

# Emory University Online Consent to Participate in Survey and ASCENT Project to Improve Kidney Transplant Waitlisting

Study Title: Evaluation of a Systems-Level Approach to Providing Education about the Kidney Allocation Policy

<u>Principal Investigator</u>: Rachel E. Patzer, Department of Surgery, Division of Transplantation

#### **Introduction and Study Overview**

Thank you for your interest in our project aimed to provide education about the kidney allocation system and transplant. We would like to tell you everything you need to think about before you decide whether or not to join.. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the project.

The purpose of this project is to test the effectiveness of quality improvement and educational materials intended for dialysis facility medical directors, staff, and patients. If you are receiving this survey, your ESRD Network is participating in this project, and your dialysis clinic has been selected to receive educational materials regarding the new kidney allocation policy.

- 1) If you join the study, you will receive educational materials in an email from and also via mail. You will also be asked to take this survey at baseline and another follow-up survey in 3 months that asks questions regarding your knowledge about the kidney allocation system, staff training, and your intent to refer patients for kidney transplantation.
- 2) This survey should take about 10-15 minutes to complete.
- 3) The potential risks include a breach of confidentiality. The likelihood of this risk is very low as all information collected through these surveys will be kept on an encrypted computer and server. Your ESRD Network will not have access to the information you provide.
- 4) This project may benefit you by providing you, your staff, and your patients with education regarding the new kidney allocation system. If the study does not benefit you directly, we hope that what we learn from this project will benefit patients and providers in the future by learning what educational materials improve access to the kidney transplant waitlist.
- 5) You will be offered a \$10 gift card for your time if you complete the baseline survey. In 3 months, you will receive \$10 again for completing the follow-up survey.
- **6)** Your privacy is very important to us.
- 7) The only protected health information we will be asking to collect from you during these surveys is your email. Providing your email is optional, and we will only be collecting this information to send you a gift card and will not share this information.
- 8) The following persons or groups may use and /or disclose your information for this project:
  - The Principal Investigator and the research staff.
- 9) Since the project data will not be linked to your name or protected health information, other people or organizations may be able to use data from this study, though we do not plan to share it.
- **10)** You may revoke your authorization at any time by calling the Principal Investigator, Rachel E. Patzer.

#### **Contact Information**

If you have questions about this project, your part in it, your rights as a participant, or if you have questions, concerns or complaints about the research you may contact the following:

| Dr. Rachel E. Patzer, Principal Investigator | : |
|----------------------------------------------|---|
| Emory Institutional Review Board: | |

## Consent

By clicking here, I consent and wish to enter the study